CLINICAL TRIAL: NCT04976413
Title: Efficacy of Eye Movement Desensitization and Reprocessing (EMDR) Psychotherapy in the Treatment of Depression and Comorbid Anxiety: A Randomized Control Trial
Brief Title: Efficacy of EMDR in the Treatment of Depression and Comorbid Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Quaid-e-Azam University (Other)
Responsible Party: Principal Investigator, Yasmeen Wajid Mauna Gauhar, Principal Investigator, Quaid-e-Azam University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB: F.No. D-107-1(03)
Record Dates: First submitted 2021-06-22; First posted 2021-07-26 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2021-07

CONDITIONS: Depression; Anxiety
Keywords: EMDR; depression; anxiety; RCT
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Eye Movement Desensitization Reprocessing; Psychotherapy; Counseling

STUDY DESIGN:
Intervention Model Description: Randomized Control Clinical Trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessment and assignment to experimental and control conditions will be carried out by an independent evaluator who will be blind to the research hypotheses; treatment providers will be blind to the scores of participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Experimental arm will receive eight phase EMDR treatment using standard protocol. Selection of targets for reprocessing through EMDR will be made according to adaptive information processing model's postulations, that links traumatic events with the symptoms of depression and anxiety. Time period allocated to EMDR treatment is 12 -14 weeks . Follow up will be conducted after 12 weeks of treatment completion.
  Interventions: Behavioral: Eye Movement Desensitization and Reprocessing (EMDR) psychotherapy
- Control (Active Comparator): Control group will receive treatment as usual (supportive counselling) for 12 -14 weeks
  Interventions: Behavioral: Counselling as usual

INTERVENTIONS:
Behavioral: Eye Movement Desensitization and Reprocessing (EMDR) psychotherapy — Experimental arm will receive eight phase EMDR treatment using manualized standard protocol. Selection of targets for reprocessing through EMDR will be made according to adaptive information processing model's postulations, that links traumatic events with the symptoms of depression and anxiety. Time period allocated to EMDR treatment is 12-14 weeks.
  Other Names: EMDR
  Arms: Experimental
Behavioral: Counselling as usual — Control arm will receive counseling as usual for 12-14 weeks
  Arms: Control

SUMMARY:
This research is aimed at investigating the efficacy of eye movement desensitization and reprocessing (EMDR) psychotherapy for treating depression and comorbid anxiety symptoms. EMDR has been scientifically established as an evidenced based level-A treatment for PTSD. However, researchers have started assessing its efficacy for depression and other psychological disorders. Preliminary evidence indicates that EMDR has the potential to treat depression, however, it has not yet been established as an evidence-based intervention. Anxiety most often comorbid with depression. literature suggests that when depression is treated, the comorbid anxiety symptoms are also reduced. Hence, the effect of EMDR therapy on anxiety symptoms, when treating depressive symptoms would also be explored.

A sample of 40 volunteers will be sought from community through advertising, and through referrals and will be randomly assigned to experimental and control conditions. Participants of experimental condition will be offered eight phase EMDR therapy in a period of 12-14 weeks. Participants of control group will receive counselling as usual sessions for 12-14 weeks. Measurement of the depression and anxiety symptoms for Experimental group will be recorded at Time 1, (baseline, time frame: 0 week). Time 2 (after history and preparation for EMDR, time frame: 3 weeks). Time 3, (after EMDR treatment, time frame: 12 weeks) and at T4, ( post treatment follow-up, Time frame: 24 weeks. For Control group, measurements will be recorded at T1, T2 and T3.

The current study will be the first registered Randomized Control Trial (RCT ) as per investigators knowledge, that will explore the efficacy of EMDR in treating depression and comorbid anxiety. The results of the study will provide the scientific bases to use EMDR as a treatment of choice for depression and anxiety. Many clients do not respond to pharmacological as well other psychological treatments despite bearing huge financial cost. EMDR therapy can be a short-term treatment that may provide relief from symptoms of depression and anxiety, and as a result, the functioning and quality of life of the participants will also improve. This study will also guide further research to explore the effects of EMDR on other trauma-based disorders and comorbid conditions.

DETAILED DESCRIPTION:
Depression is the foremost cause of global disease and disability burden . It often coexists with other chronic diseases and exacerbates health related outcomes . The prevalence rate of depression and anxiety is on the rise in Pakistan due to various challenging conditions . Hence, there is a greater need to find new and effective treatment/s, that would supplement the existing treatments in treating depression and anxiety.

Depression is usually treated through antidepressants, counselling or psychotherapy. However, antidepressants have shown a meek advantage over placebos, and its use increases with rise in the severity of depression. Therefore, pharmacological treatment should only be opted for if depression is moderate to severe and does not respond to psychotherapy; or when psychotherapy is not available . Cognitive Behavioral Therapy (CBT) is the recommended therapy to treat depression . It significantly reduces relapse rate occurrence . A meta-analysis of 28 studies found CBT effective in reducing the relapse rate significantly for Major Depression compared to pharmacotherapy . On the contrary, the meta-analysis of 70 studies reported a linear and steady decline in the effectiveness of CBT across time with contemporary CBT seemingly providing less relief from depressive symptoms as compared to its effectiveness reported in previous years. EMDR therapy has also been researched to treat depression. Preliminary evidence exists through case studies and limited research that EMDR has the potential to treat trauma induced depressive symptoms.

Comorbidity of Depression and Anxiety: Anxiety and depression occupy top ten of leading causes of global disease burden . World Health Organization estimated that 4.4% of the global population was living with depression and 3.6% was suffering from an anxiety disorder. Generalized anxiety, social anxiety, and depression comorbid substantially and pervasively with depression . It leads to impaired functioning and requires additional treatment . The depression anxiety co-occurrence was also found to be significant across developmental periods, and the relationship between the two disorders was linked to stressful events experienced in childhood.

The prevalence rate of depression and anxiety in various localities in Pakistan ranges from 22% to 60 %, which is very high compared to other developing countries . Hence, it is a significant mental health concern requires serious attention. Hence, EMDR efficacy to treat depression and comorbid anxiety is explored through this study. According to a meta-analysis, psychotherapy targeted at treating depression can also decrease anxiety symptoms compared to control conditions.

Eye Movement Desensitization and Reprocessing (EMDR) is scientifically validated and an integrative psychotherapeutic intervention which was initially introduced as a treatment for post-traumatic stress disorder (PTSD). There is a strong research support for EMDR efficacy in treating PTSD and comorbid conditions. literature suggested EMDR as a positive treatment for depression . A meta-analysis on treatment of PTSD and depression showed that EMDR seems to have significantly stronger effect on comorbid depression than CBT. However, research in this regard is scant. Studies conducted so far suggests that EMDR has a greater potential to treat depression and anxiety . An unpublished pilot study (N=16) conducted earlier by this researcher has provided preliminary support for this assumption. The current study will investigate the effect of EMDR therapy on depression and comorbid anxiety symptoms on a sample of 40 participants.

Research Questions: Is EMDR an effective intervention for treating depression? Can EMDR also reduce comorbid anxiety symptoms in depressed individuals? Will the quality of life and functioning of the participants improve after amelioration of depressive and anxiety symptoms? Objectives: The objectives are to assess the efficacy of EMDR in treating individuals with depression, analyze EMDR's impact on comorbid anxiety symptoms and find the effects of EMDR on the quality of life and functioning of the participants.

Hypotheses: (1) There will be significant reduction in the depressive symptoms of the experimental participants after treatment as compared to symptoms reported before treatment. (2) There will be significant reduction in comorbid anxiety symptoms of experimental participants after treatment as compared to symptoms reported before treatment. (3) The quality of life and functioning of experimental participants will improve after EMDR treatment as compared to quality of life and functioning reported before treatment. (4) There will be significant reduction in the depressive symptoms of experimental group participants after treatment compared to depressive symptoms of control group participants. (5) There will be significant reduction in comorbid anxiety symptoms of experimental group after treatment compared to the symptoms reported by the control group participants.

Procedure: Participants' selection will be based on inclusion criteria assessed through clinical interview, scores on research instruments and signing of the informed consent. Assessment and random assignment to an experimental and a control condition will be carried out by an independent assessor who will be blind to the research hypotheses. The baseline assessment will be conducted at T1 i.e Week 0. The second assessment T2, will be carried out after 3 weeks for both the groups. During these 3 weeks experimental group participants will provide history, learn safe place and other grounding techniques, and select targets for EMDR treatment. The control group will carry on with treatment as usual. For the next 6-9 weeks both the groups will receive their respective treatments. Third assessment (T3) will be carried out after treatment completion for both the groups at week 12 . Experimental group participants will have a follow-up assessment (T4) after week 24.

Statistical analysis of Paired and Independent t-test would evaluate EMDR treatment effects within and between groups. Results would be discussed and published after the study is completed.

ELIGIBILITY:
Inclusion Criteria:

* 18-item Clinically Useful Depression Outcome Scale (CUDOS) scores of 20 or more;
* 20-item Clinically Useful Anxiety Outcome Scale (CUXOS) scores of 20 or more;
* IES scores of less than or equal to 33
* DES scores of less than or equal to 36
* English or Urdu speaking
* Ability to understand terms and willingness to participate in the study, give informed consent
* Currently not taking any psychological or psychiatric treatment
* No substance dependence (except tobacco smoking)

Exclusion Criteria:

* Brain injury/ organicity, neurological illnesses, high dissociation, PTSD
* Schizophrenia/ psychotic disorders spectrum
* Bipolar disorders
* Substance dependence
* Other disorders poorly suited to study treatments (e.g., personality disorders)
* Serious suicidal ideation that requires immediate attention
* Any psychiatric or medical condition impeding participation in the study
* Current pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
DSM-5 Self-Rated Level 1 Cross Cutting Symptoms Measure Adult, English and Urdu versions | Week 0, baseline
  Measures cross cutting symptoms across psychiatric domains. Scores on each item ranges from 0-4. A score of 0 indicates no symptoms and 4 means worst outcome
Clinically Useful Depression Outcome Scale, English and Urdu versions | week 0, week -3, week 12, week 24
  Measures baseline and changes in depressive symptoms, functioning and quality of life, scores on each item ranges from 0-4. A score of 0 indicate no symptoms and 4 means worst outcome
Clinically Useful Anxiety Outcome Scale, English and Urdu versions | week 0, week -3, week 12, week 24
  Measures baseline and changes in anxiety symptoms, scores on each item ranges from 0-4. A score of 0 indicates no symptoms and 4 means worst outcome
Dissociative Experience Scale-II, English and Urdu versions | Week 0,
  Measures dissociative symptoms scores on each item ranges from 0%-100%. A score of 0% indicates no symptoms and 100% means worst outcome
Impact of Event scale, English and Urdu versions | Week 0,
  Measures event-specific distress, scores on each item ranges from 0-4. A score of 0 indicates no symptoms and 4 means worst outcome

CONTACTS AND LOCATIONS:
Overall Officials: Yasmeen W Mauna Gauhar, M.Phil, Principal Investigator — National Institute of Psychology, Quaid i Azam University Islamabad Pakistan; Dr. Humaira Jami, Ph.D, Study Chair — National Institute of Psychology, Quaid i Azam University Islamabad Pakistan; Dr Derek Ferrel, Ph.D, Study Chair — University of Worcester. U.K.; Dr Wajid Malik, MBBS FCPS, Study Director — Armed Forces Institute of Mental Health, Rawalpindi Pakistan
Locations (2):
- Pakistan (2):
  - Growing Edge Consultants, Islamabad, Federal Territory
  - National Institute of Psychology, Center of Excellence, Quaid i Azam University, Islamabad, Pakistan., Islamabad, Federal Territory

IPD SHARING:
Plan to Share IPD: No
Individual participant data dictionaries (IDP) will not be shared with other researchers in future. The current study is based on a pilot study conducted earlier. Participants of the pilot study did not agreed to share their IDP in the past. The decision for not sharing IDP is based on having consideration for the participants informed consent which may be influenced by their culture. However, study protocol, statistical analysis plan, informed consent form to participate in the study and clinical study report will be available for viewing after the study is completed.